CLINICAL TRIAL: NCT02726711
Title: Reduction in Splanchnic Capacitance Contributes to Sympathetically Dependent Hypertension in Autonomic Aim 1 of Rare Diseases Clinical Research Network (RDCRN) Project 2
Brief Title: Reduction in Splanchnic Capacitance Contributes to Sympathetically Dependent Hypertension in Autonomic
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, MD, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 151947
Record Dates: First submitted 2016-01-28; First posted 2016-04-04 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Multiple System Atrophy; Orthostatic Hypotension; Supine Hypertension
MeSH Terms: conditions — Multiple System Atrophy; Hypotension, Orthostatic | interventions — Trimethaphan; trimethaphan camsylate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trimethaphan (Experimental): The investigator will measure cardiac output by studying the air the participant breathes in and out. The participant will also wear a facemask to apply a low air pressure to the airway.
  After this, the trimethaphan infusion will begin with a small dose and the investigators increase at 1-2 minute intervals for up to five doses. The measurements will be collected again.
  Next, a standard blood pressure cuffs will be wrapped around the participant's abdomen. the cuff will inflate to apply pressure for 5 - 15 minutes.
  Interventions: Drug: Trimethaphan
- Placebo (Placebo Comparator): The investigator will measure cardiac output by studying the air the participant breathes in and out. The participant will also wear a facemask to apply a low air pressure to the airway.
  After this, the placebo (saline) infusion will begin with a small dose and the investigators increase at 1-2 minute intervals for up to five doses. The measurements will be collected again.
  Next, a standard blood pressure cuffs will be wrapped around the participant's abdomen. the cuff will inflate to apply pressure for 5 - 15 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trimethaphan — Trimethaphan will be infused (0.5 - 4.0 mg IV)
  Other Names: Trimethaphan Camsylate
  Arms: Trimethaphan
Drug: Placebo — 0.5 - 4.0 mg IV to be infused
  Other Names: saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn more about the regulation of the veins of the abdomen by the autonomic (involuntary) nervous system, and how this may affect high blood pressure. Normally, the autonomic nervous system controls how much blood flows in the veins. In people with high blood pressure, however, the autonomic nervous system is changed. This change may affect the way blood flows in the veins of the abdomen which may play a role in their high blood pressure. About 32 participants will be screened for the study. The investigators estimate 16 will be eligible to participate in all of the study days.

DETAILED DESCRIPTION:
The investigators will study male and female subjects, age 40-80 years with possible or probable Multiple System Atrophy, as defined by Consensus Criteria who suffer from supine hypertension defined as SBP≥150, and neurogenic orthostatic hypotension, defined as a ≥30-mmHg decrease in systolic BP within 3 minutes of standing associated with impaired autonomic reflexes determined by autonomic testing in the absence of other identifiable causes. All participants will be able and willing to provide informed consent.

Screening Procedures. Potential participants will be studied in the Vanderbilt Autonomic Dysfunction Center (ADC). Medications affecting BP, blood volume and the autonomic nervous system such as antihypertensives, pressor medications and fludrocortisone will be withdrawn for at least 5 half-lives before studies. Screening procedures can be performed in one or more days depending on the patient's and investigator's availability.

* Patients will undergo a complete history and physical examination, ECG, routine clinical laboratory analysis and a blood pregnancy test for women with childbearing potential.
* Autonomic testing including sinus arrhythmia, Valsalva maneuver and a posture study with plasma catecholamines is then performed to determine if they meet the inclusion/exclusion criteria. During these tests, blood pressure (BP) and heart rate (HR) will be obtained using an automated oscillometric sphygmomanometer, finger photoplethysmography, and continuous ECG. During the orthostatic test, blood samples will be obtained for hormones that regulate BP, such as catecholamines, while patients are supine and upright.

Medical history information and results from any of the screening procedures obtained within the previous 6 months for other studies within this research group may be utilized.

Study Procedures: Study Day 1 and 2

Eligible Multiple System Atrophy patients with supine hypertension will be studied twice in a randomized, single blind, crossover design, once with trimethaphan and once with placebo. The order of administration is randomized. The placebo day will have identical interventions, but saline will be infused instead of trimethaphan to provide a time control. Studies will be conducted in a postvoid state and ≥2 hours after meals. Each study day will last 2-3 hours. The following procedures will be conducted:

Patients will be instrumented to measure blood pressure continuously with photoplethysmography, and intermittently with an automated oscillometric device. Heart rate will be monitored continuously with ECG. Electrodes will be placed on thorax and abdomen to measure segmental impedance. Skin blood flow will be measured in the forearm with a laser Doppler. Cardiac output will be measured by the inert gas rebreathing technique and/or by impedance cardiography. An IV will be placed in one arm for drug administration.

After instrumentation baseline measurements will be recorded, including cardiac output and splanchnic venous capacitance. Venous capacitance will be estimated using an adaptation of the method of Schmitt et al. In this technique, segmental impedance is monitored, while continuous positive airway pressure (CPAP) is applied sequentially at 0, 4, 8, 12 and 16 cm water (H20) for 1-2 minute each.

Patients will then receive either placebo (time control) or trimethaphan, to induce complete withdrawal of residual sympathetic tone. Intravenous infusion of trimethaphan camsylate (Cambridge Labs) will be started at 0.5-1 mg/min and increased by 1.0 mg/min in 2-6 minute intervals to one of the following endpoints: presyncopal symptoms, no further decrease in blood pressure with increased infusion rates, or an infusion rate of 4 mg/min. Once a stable decrease in blood pressure is obtained, outcome measurements will be repeated.

Abdominal compression will be applied to a sustained 40 mm Hg pressure while supine with an inflatable binder. Outcome measurements will be repeated 5-15 minutes later. The investigator may decide not to perform this procedure (due to a longer than anticipated study day duration / drug infusion). In this case, the study will include only the outcome measurements during the drug infusion.

The infusion of trimethaphan is then stopped and patient monitored until blood pressure is restored to baseline values.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age 40-80 years, with possible or probable Multiple System Atrophy, as defined by Consensus Criteria.
* Neurogenic orthostatic hypotension defined as a ≥30-mmHg decrease in systolic blood pressure within 3 minutes of standing associated with impaired autonomic reflexes determined by autonomic testing in the absence of other identifiable causes.
* Supine hypertension, defined as systolic blood pressure ≥150 mmHg measured on two separate occasions.
* Subjects able and willing to provide informed consent.

Exclusion Criteria:

* Pregnancy.
* Systemic illnesses known to produce autonomic neuropathy, including but not limited to diabetes mellitus, amyloidosis, monoclonal gammopathies, and autoimmune neuropathies
* History of known aortic aneurysms, thoracic, abdominal or pelvic surgery in the past 6 months
* Symptomatic abdominal or inguinal hernias
* Severe gastroesophageal reflux
* Recent fractures or fissures of ribs, thoracic or lumbar spine
* Medical devices implanted on the abdominal wall or abdomen that would interfere with the abdominal compression
* Intolerance to any increase in intra-abdominal pressure
* Clinically unstable coronary artery disease or major cardiovascular or neurological event in the past 6 months, and other factors which in the investigator's opinion would prevent the subject from completing the protocol including clinically significant abnormalities in clinical, mental or laboratory testing.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-04; Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The percentage of increase of the y intercept of the P-V relationship | 5 years
  To determine whether autonomic blockade with trimethaphan increases splanchnic capacitance (parallel upward shift in the P-V relationship) compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No